CLINICAL TRIAL: NCT05266664
Title: Preterm Immune System Development and Response to Immunization
Acronym: PRIMI
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Amphia Hospital (Other); Albert Schweitzer Hospital (Other); Franciscus Gasthuis (Other); Maasstad Hospital (Other); Maxima Medical Center (Other); Reinier de Graaf Groep (Other); Erasmus Medical Center (Other); Merck Sharp & Dohme LLC (Industry); Zuyderland Medical Centre (Other); Haga Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL80118.068.22
Record Dates: First submitted 2022-02-11; First posted 2022-03-04 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Immune System Disorder; Preterm; Vaccination Failure
Keywords: immune system development; preterm infant; vaccination
MeSH Terms: conditions — Immune System Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white blood cells, stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm: preterm infants gestational age less than 32 weeks
- healthy controls: healthy term infants

SUMMARY:
In this study the response to vaccination and development of the immune system in very preterm infants upon the current vaccination schedule will be compared to healthy term infants.

DETAILED DESCRIPTION:
Preterm infants are at increased risk of developing infections early in life due to a less mature immune system compared to full-term infants. Moreover, protection by the placental transfer of maternal antibodies in general and specifically against vaccine antigens has shown to be significantly lower in very preterm infants (gestational age (GA)< 32 weeks) compared to term infants. In this study we aim to investigate the immune system development of very preterm infants. Adequate immune response to vaccination is considered both clinically important as well as a functional test of the immune system. However, data on the antibody and Ag-specific memory B cell response to vaccination in preterm infants are limited.

Primary objective is to study the antibody immune response to routine vaccinations in very preterm infants (GA<32 weeks). Secondary aim is to study the immune system more extensively using flow cytometry, ELISA and single cell transcriptomics to measure development of Ag-specific memory B cells raised in response to vaccination, and by using proteomics, epigenetics, and microbiome studies.

ELIGIBILITY:
To be eligible to participate in this study, a preterm infant must meet all following criteria:

* Preterm infant born at gestational age less than 32 weeks (whose mothers did or did not receive a T dap vaccination during pregnancy)
* Parents/ guardians must have sufficient understanding of the Dutch language

To be eligible to participate in this study, a healthy full-term infant must meet all following criteria:

* healthy full-term infant whose mother received a Tdap vaccination during pregnancy
* Parents/ guardians must have sufficient understanding of the Dutch language

To be eligible to participate in this study, a mother must meet all following criteria:

- Mother of preterm or health full-term infant who are participating in the study

Exclusion Criteria:

* Parents/guardians of the infant are not able or willing to provide informed consent
* Infant with congenital anomaly which are more likely to cause adverse effects after immunization (for example hemodynamically significant congenital heart defect)
* Infant with a (possible) HIV infection or immunodeficiency
* Maternal use of immunosuppressive drugs during pregnancy

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For this study 120 preterm infants (GA< 32 weeks) and their mothers will be enrolled to evaluate the antibody response to vaccination and the development of the immune system. In a subgroup of 25 preterm infants after maternal Tdap vaccination and 25 preterm infants whose mothers did not receive Tdap vaccination, Ag-specific memory B cell response to vaccination will be studied. For comparison of Ag-specific memory B cell development 25 healthy term infants and their mothers will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
antibody immune response to routine vaccinations in very preterm infants | 6 months
  IgG antibody concentrations against six vaccine antigens in preterm-born infants following primary series of routine vaccinations with Vaxelis in order to assess the proportion of children with IgG concentrations above international-defined thresholds for protection.

SECONDARY OUTCOMES:
IgG antibody concentrations following booster of routine vaccination with Vaxelis | 12 months
  IgG antibody concentrations against vaccine antigens in preterm-born infants following booster of routine vaccination with Vaxelis.
geometrical mean concentrations following primary series and booster of routine vaccination with Vaxelis. | 6 and 12 months
  geometrical mean concentrations in preterm infants compared to reference values in healthy term infants as known from literature following primary series and booster of routine vaccination with Vaxelis.
IgG antibody concentrations following routine vaccinations with 10-valent pneumococcal conjugate vaccine after primary series and booster vaccination. | 6 and 12 months
  IgG antibody concentrations against vaccine antigens in preterm-born infants following routine vaccinations with 10-valent pneumococcal conjugate vaccine after primary series and booster vaccination.
IgG antibody concentrations against pertussis antigens at 2 months of age in preterm-born infants after maternal Tdap vaccination and in infants whose mother did not receive maternal Tdap vaccination. | 2 months
  IgG antibody concentrations against pertussis antigens at 2 months of age (before start of infant immunizations) in preterm-born infants after maternal Tdap vaccination and in infants whose mother did not receive maternal Tdap vaccination.
number of antigen-specific memory B cells in cells/microliter following routine vaccinations after primary series and booster vaccination | 6 and 12 months
  number of antigen-specific memory B cells in cells/microliter in preterm-born infants following routine vaccinations after primary series and booster vaccination
IgG antibody concentrations in relation to maternal antibody concentrations against vaccine antigens | birth, 2,6 and 12 months
  IgG antibody concentrations against vaccine antigens in preterm-born infants before start of immunizations and following routine vaccinations after primary series and booster vaccination, in relation to maternal antibody concentrations against vaccine antigens
comparison of response to vaccination between preterm infants and healthy term infants | 6 and 12 months
  Proportions of infants with IgG concentrations above the internationally defined threshold for protection and geometrical mean concentrations will be compared between preterm infants after maternal Tdap vaccination, preterm infants whose mothers did not receive Tdap vaccination and reference values in healthy term infants as known from literature.
Comparison of number of antigen-specific memory B cells in cells/microliter with and without preceding maternal Tdap vaccination | 6 and 12 months
  Number of antigen-specific memory B cells in cells/microliter will be compared between preterm infants after maternal Tdap vaccination, preterm infants whose mothers did not receive Tdap vaccination and healthy term infants after maternal Tdap vaccination, who will be recruited for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Driessen, Prof MD PhD, Study Director — Maastricht UMC; Jantien Bolt-Wieringa, MD, Principal Investigator — Medical Center Haaglanden
Locations (7):
- Netherlands (7):
  - Amphia Hospital, Breda
  - reinier de Graaff Group, Delft
  - Albert Schweitzer Hospital, Dordrecht
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Maxima Medical Center, Veldhoven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collins A, Weitkamp JH, Wynn JL. Why are preterm newborns at increased risk of infection? Arch Dis Child Fetal Neonatal Ed. 2018 Jul;103(4):F391-F394. doi: 10.1136/archdischild-2017-313595. Epub 2018 Jan 30. PMID 29382648
- [Background] Heininger U, Riffelmann M, Leineweber B, Wirsing von Koenig CH. Maternally derived antibodies against Bordetella pertussis antigens pertussis toxin and filamentous hemagglutinin in preterm and full term newborns. Pediatr Infect Dis J. 2009 May;28(5):443-5. doi: 10.1097/INF.0b013e318193ead7. PMID 19319020
- [Background] van den Berg JP, Westerbeek EA, Berbers GA, van Gageldonk PG, van der Klis FR, van Elburg RM. Transplacental transport of IgG antibodies specific for pertussis, diphtheria, tetanus, haemophilus influenzae type b, and Neisseria meningitidis serogroup C is lower in preterm compared with term infants. Pediatr Infect Dis J. 2010 Sep;29(9):801-5. doi: 10.1097/inf.0b013e3181dc4f77. PMID 20803841
- [Background] Wilck MB, Xu ZJ, Stek JE, Lee AW. Safety and immunogenicity of a fully-liquid DTaP-IPV-Hib-HepB vaccine (Vaxelis) in premature infants. Hum Vaccin Immunother. 2021 Jan 2;17(1):191-196. doi: 10.1080/21645515.2020.1756668. Epub 2020 Aug 4. PMID 32750261
- [Background] Barug D, Pronk I, van Houten MA, Versteegh FGA, Knol MJ, van de Kassteele J, Berbers GAM, Sanders EAM, Rots NY. Maternal pertussis vaccination and its effects on the immune response of infants aged up to 12 months in the Netherlands: an open-label, parallel, randomised controlled trial. Lancet Infect Dis. 2019 Apr;19(4):392-401. doi: 10.1016/S1473-3099(18)30717-5. Epub 2019 Mar 27. PMID 30938299
- [Background] Syed YY. DTaP5-HB-IPV-Hib Vaccine (Vaxelis(R)): A Review of its Use in Primary and Booster Vaccination. Paediatr Drugs. 2017 Feb;19(1):69-80. doi: 10.1007/s40272-016-0208-y. PMID 28035545
- [Background] Vono M, Eberhardt CS, Auderset F, Mastelic-Gavillet B, Lemeille S, Christensen D, Andersen P, Lambert PH, Siegrist CA. Maternal Antibodies Inhibit Neonatal and Infant Responses to Vaccination by Shaping the Early-Life B Cell Repertoire within Germinal Centers. Cell Rep. 2019 Aug 13;28(7):1773-1784.e5. doi: 10.1016/j.celrep.2019.07.047. PMID 31412246